CLINICAL TRIAL: NCT03963882
Title: Neoadjuvant Chemotherapy Followed by Radical Hysterectomy for the Treatment of Locally Advanced Cervical Cancer: A Prospective Cohort Study
Brief Title: NAC Followed by RH for the Treatment of LACC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACC
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Neoadjuvant Chemotherapy; Locally Advanced Cervical Cancer; Radical Hysterectomy; Objective Response; Laparoscopy; Laparotomy; Concurrent Chemoradiotherapy; Adjuvant Therapy; Systematic Chemotherapy
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: patients diagnosed with locally advanced cervical cancer of stage IB2 to IIB (FIGO 2009 system)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Patients in group A don't receive neoadjuvant chemotherapy
  Interventions: Diagnostic Test: First imaging evaluation; Radiation: Radiochemotherapy
- Group B (Experimental): Patients in group B receive neoadjuvant chemotherapy and achieve imaging response
  Interventions: Drug: Two cycles of neoadjuvant chemotherapy; Diagnostic Test: First imaging evaluation; Diagnostic Test: Second imaging evaluation; Drug: The third cycles of neoadjuvant chemotherapy; Procedure: RH; Diagnostic Test: Pathologic evaluation
- Group C (Experimental): Patients in group B receive neoadjuvant chemotherapy but don't achieve imaging response, and they accept concurrent chemoradiotherapy
  Interventions: Drug: Two cycles of neoadjuvant chemotherapy; Diagnostic Test: First imaging evaluation; Diagnostic Test: Second imaging evaluation; Radiation: Radiochemotherapy
- Group D (Experimental): Patients in group B receive neoadjuvant chemotherapy but don't achieve imaging response, and they accept radical hysterectomy
  Interventions: Drug: Two cycles of neoadjuvant chemotherapy; Diagnostic Test: First imaging evaluation; Diagnostic Test: Second imaging evaluation; Procedure: RH; Diagnostic Test: Pathologic evaluation

INTERVENTIONS:
Drug: Two cycles of neoadjuvant chemotherapy — Two cycles of neoadjuvant chemotherapy (paclitaxel 175 mg/m2 and cisplatin 70 mg/m2, on day 1, once for three weeks).
  Arms: Group B; Group C; Group D
Diagnostic Test: First imaging evaluation — First imaging evaluation consists of pelvic magnetic resonance imaging (MRI) and positron emission tomography (PET)
Diagnostic Test: Second imaging evaluation — Second imaging evaluation consists of pelvic magnetic resonance imaging
  Arms: Group B; Group C; Group D
Drug: The third cycles of neoadjuvant chemotherapy — The third cycles of neoadjuvant chemotherapy (paclitaxel 175 mg/m2 and cisplatin 70 mg/m2, on day 1, once for three weeks).
  Arms: Group B
Procedure: RH — Radical hysterectomy
  Arms: Group B; Group D
Radiation: Radiochemotherapy — Concurrent radiochemotherapy
  Arms: Group A; Group C
Diagnostic Test: Pathologic evaluation — Pathologic evaluation for RH patients
  Arms: Group B; Group D

SUMMARY:
This cohort study is to evaluate the role of neoadjuvant chemotherapy (NAC) in the treatment of locally advanced cervical cancer (LACC). Sixty patients with LACC (FIGO 2009 stage IB2 to IIB) will be enrolled. After informed consents, they would accept the imaging evaluation of pelvic magnetic resonance imaging (MRI) and positron emission tomography (PET). After excluding cases of distant metastasis, they will accept two cycles of NAC (paclitaxel 175 mg/m2 and cisplatin 70 mg/m2, on day 1, once for three weeks). Then a second MRI is performed to evaluate the imaging response. For patients achieving objective response, radical hysterectomy (RH, via laparoscopy or laparotomy) and an evaluation of pathologic response are performed. For patients without objective imaging response, the choice of concurrent chemoradiotherapy or radical hysterectomy will be discussed. After RH, adjuvant therapy will be given according to the RH pathologic results.

The primary objectives consist of (1) the objective imaging response after NAC; (2) the objective pathologic response after RH.

The secondary objectives consist of (1) disease-free survival and overall survival after various therapy modalities; (2) severe adverse effects of NAC; (3) the effects of NAC on the surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix
* FIGO stage IB2 to IIB
* Type II or III radical hysterectomy or trachelectomy
* Performance status of Eastern Cooperative Oncology Group (ECOG) 0-1
* Aged 18 years to 45 years
* Well cardiopulmonary, liver and kidney functions for neoadjuvant chemotherapy
* Signed an approved informed consents

Exclusion Criteria:

* Not satisfying any of the inclusion criteria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective pathologic response | 3 years
  Objective pathologic response for patients with radical hysterectomy
Objective imaging response | 3 years
  Objective imaging response for patients with neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  Disease-free survival for patients with various therapy modalities
Overall survival | 3 years
  Overall survival for patients with various therapy modalities
Severe adverse events | 1 year
  Severe adverse events of neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No